CLINICAL TRIAL: NCT06204796
Title: The Role of Vitamin D in Amelioration of Oral Lichen Planus and Its Effect on Salivary IFN-γ Level: a Randomized Clinical Trial
Brief Title: The Role of Vitamin D in Amelioration of Oral Lichen Planus and Its Effect on Salivary IFN-γ Level
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Fayoum University (Other)
Responsible Party: Principal Investigator, Rania Hassan Shalby, Lecturer of Oral Medicine, Fayoum University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 19038219038211013
Record Dates: First submitted 2023-09-10; First posted 2024-01-12 (Actual); Last update posted 2024-01-12 (Actual); Status verified 2024-01

CONDITIONS: Oral Lichen Planus; Vitamin D Deficiency
Keywords: vitamin D, Oral Lichen Planus, salivary IFN-γ
MeSH Terms: conditions — Lichen Planus, Oral; Vitamin D Deficiency

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vitamin D+ Systemic steroids (Active Comparator): vitamin D supplement was given as 60,000 IU weekly in conjunction with systemic steroids.
  Interventions: Drug: vitamin D supplement was given as 60,000 IU weekly in conjunction with systemic prednisone; Drug: Systemic prednisone
- Systemic steroids alone (Active Comparator): systemic steroids only
  Interventions: Drug: Systemic prednisone

INTERVENTIONS:
Drug: vitamin D supplement was given as 60,000 IU weekly in conjunction with systemic prednisone — All participants received 40-60 mg of systemic prednisone as a single morning dose according to the severity of the condition until a 50% reduction in lesion size was achieved then the dose was tapered by 10mg each week and finally to 5 mg/day for the last week. Patients were followed up weekly for up to 60 days. The length and dose of treatment were adjusted according to clinical needs in each case. In addition, a vitamin D supplement was given as 60,000 IU weekly in conjunction with systemic steroids.
  Arms: Vitamin D+ Systemic steroids
Drug: Systemic prednisone — All participants received 40-60 mg of systemic prednisone as a single morning dose according to the severity of the condition until a 50% reduction in lesion size was achieved then the dose was tapered by 10mg each week and finally to 5 mg/day for the last week. Patients were followed up weekly for up to 60 days. The length and dose of treatment were adjusted according to clinical needs in each case.

SUMMARY:
The goal of this clinical trial is to compare between the use of vitamin D supplement in conjunction with systemic steroids versus the use of systemic steroids alone in the management of patients with symptomatic Oral Lichen Planus lesions and the comparison of salivary Interferon gamma levels in both study groups before and after treatment

DETAILED DESCRIPTION:
The objective of the research:

To investigate the role of vitamin D supplements in the management of vitamin D deficient oral lichen planus (OLP) patients and to examine its suppressive effect on pro-inflammatory cytokine (IFN-γ) in saliva samples of OLP patients

• Steps in short

1- Trial design: This study is a randomized clinical trial (RCT) having parallel groups with a 1:1 allocation ratio. This study will conform with the Consolidated Standards of Reporting Trials guidelines (CONSORT guidelines).

Middle-aged patients presenting with clinical and histopathological features of symptomatic (atrophic, erosive, or bullous) OLP (32) and having vitamin D deficiency or insufficiency (≤30 ng/ml) (33) will be included in the present study.

4-Intervention and study groups A total of 40 participants will be randomly and equally allocated into one of the two study groups to receive either, systemic steroids and vitamin D supplement (intervention) or systemic steroids only (control).

Clinical evaluation of the lesion through two components including objective morphological signs and subjective symptoms that describe the pain and burning sensation; will be measured at baseline and after 4 weeks of treatment

* Subjective findings (symptoms) using VAS score or burning sensation and pain ranging from 0 to 10 Changes in salivary INF-γ level (pg/mL) at baseline and after 4 weeks of treatment (measured using ELIZA technique)
* Treatment administration All participants will receive 40-60 mg of systemic prednisone as a single morning dose according to the severity. in the intervention group, a vitamin D supplement will be given as 60,000 IU weekly in conjunction with systemic steroids.

For the measurement of vitamin D3, The enzyme-linked immunosorbent assay (ELISA) will be used to process all samples simultaneously. Vitamin D levels lower than 30 ng/ml were assigned to vitamin D deficiency or insufficiency.

-Measurement of the inflammatory mediator (IFN-γ ) in saliva using (ELISA) kit After the initial diagnosis visit (during recruitment), patients will be clinically examined again for assessment of outcomes at baseline and after 1 month of treatment. Patients will be followed up for up to 60 days.

ELIGIBILITY:
Inclusion Criteria:

* Middle-aged patients
* Clinical and histopathological features of symptomatic (atrophic, erosive, or bullous) OLP
* Vitamin D deficiency or insufficiency (≤30 ng/ml)

Exclusion Criteria:

* Oral mucosal lesion other than OLP
* Suspected restoration-related reaction
* Active periodontitis
* Patients receiving any topical or systemic medication that may affect SVDL or induce a lichenoid reaction
* Patient having systemic disease based on the detailed questionnaire of the modified Cornell Medical Index

Ages: 35 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2023-08-01 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-01 (Actual)

PRIMARY OUTCOMES:
Severity of clinical presentation of the lesion | 1 months
  The severity of the clinical presentation of the lesion was calculated by multiplying (Sub-site score A) by (Severity score B) as Sub-site score A 0= no lesion
  1. evidence of lichen planus
  2. ≥50% of buccal mucosa, dorsum of the tongue, the floor of the mouth, hard palate, soft palate, or oropharynx affected Severity score B
  0= keratosis only
  1. keratosis with mild erythema (≤ 3 mm from gingival margin)
  2. marked erythema (e.g. full thickness of gingivae, extensive with atrophy or edema on non-keratinized mucosa)
  3. ulceration present Severity of clinical appearance=A*B (sub-site score* severity score)
     * Mild: 1-2
     * Moderate: 3-4
     * Severe: 5-6 Finally, the lesion was considered as persisting at follow-up if the clinical presentation score was greater than 0 where whereas a score of 0 indicated a healed lesion.
Pain and burning sensation | 1 months
  VAS score or burning sensation and pain ranging from 0 to 10
  * Mild : 0-4
  * Moderate: 5-7
  * Severe: 8-10

SECONDARY OUTCOMES:
Changes in salivary INF-γ level | 1 months
  Changes in salivary INF-γ level (pg/mL) at baseline and after 4 weeks of treatment (measured using ELIZA technique)

CONTACTS AND LOCATIONS:
Overall Officials: Rania H Shalby, Principal Investigator — Faculty of Dentistry-Fayoum University; Yasmine G Hamid, phd, Principal Investigator — Modern modern university for technology and information MTI University
Locations (1):
- Rania Hassan Shalby, Giza, Egypt

IPD SHARING:
Plan to Share IPD: No